CLINICAL TRIAL: NCT02264301
Title: The Effect of Qingkailing Injection on Corticosteroids Withdrawal Rate in Patients With Active Rheumatoid Arthritis
Brief Title: Qingkailing Injection Versus Puerarin Injection on Withdrawal Rate of Corticosteroids in Patients With Active Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chengdu PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yang Min, Ph.D, Chengdu PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QKL20140588
Record Dates: First submitted 2014-10-03; First posted 2014-10-15 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — puerarin; Qingkailing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Puerarin injection 400 mg (Active Comparator): Patients under the treatment of Puerarin injection 400 mg,daily,for 24 weeks
  Interventions: Drug: Puerarin injection 400 mg
- Qingkailing injection 40 ml (Experimental): Patients under the treatment of Qingkailing injection 40 ml,daily,for 24 weeks
  Interventions: Drug: Qingkailing injection 40 ml

INTERVENTIONS:
Drug: Puerarin injection 400 mg
  Arms: Puerarin injection 400 mg
Drug: Qingkailing injection 40 ml
  Arms: Qingkailing injection 40 ml

SUMMARY:
The purpose of this study is to evaluate the effect of Qingkailing injection versus Puerarin injection on withdrawal rate of corticosteroids in patients with active rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* with active RA
* without taking any other medication for the treatment of active RA in at least 4 last weeks
* aged from 18 to 75 years
* without conflict to the written, informed consent signed prior to the enrollment.

Exclusion Criteria:

* being included in other clinical trial within the last 4 weeks
* with abnormal liver or kidney function (more than 1 time above the high normal)
* with serious cardiovascular disease
* with hematologic disease
* being in pregnancy, lactation period or under a pregnancy plan
* with severe gastrointestinal disease
* with contraindication or being allergic to the test drugs
* being under the treatment of drugs within 1 previous week, that might affect the results of the trial, such as non-steroidal anti-inflammatory drugs, steroidal anti-inflammatory drugs, immunosuppressants, anti-ulcer drugs
* being not compatible for the trial medication, or other circumstances at the discretion of investigators
* without legal capacity or only with limited legal capacity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in corticosteroids withdrawal rate at 24 weeks | At 0 week, 12 weeks, 24 weeks
  The number (rate) of patients who do not need the use of corticosteroids any more were monitored 0 week, 12 weeks, 24 weeks.

SECONDARY OUTCOMES:
Change from baseline in Disease activity score in 28 joints(DAS28) | At 0 week, 12 weeks, 24 weeks
  Disease activity of RA is assessed using disease activity score in 28 joints (DAS28). DAS28 = 0.56 • √(tender joint count) + 0.28 •√(swollen joint count) + 0.70 In(ESR) + 0.014(global health on visual analogue scale).DAS28 will be assessed at At 0 week, 12 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Chengdu Military Area Command PLA, Chengdu, China